CLINICAL TRIAL: NCT02884830
Title: Does Nocturnal Continuous Positive Airway Pressure Use Improves Sleep Quality in Chronic Obstructive Pulmonary Disease Patients?
Brief Title: Nocturnal Continuous Positive Airway Pressure in Chronic Obstructive Pulmonary Disease Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: the protocol is too complex and we are not able to recruit appropriate patients
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK/16-05-73/4668AD
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham CPAP (Placebo Comparator): Sham continuous positive airway pressure is a CPAP given at too low pressure to have any physiological effect on upper airways patency and on lung volumes
  Interventions: Device: continuous positive airway pressure
- Efficace CPAP (Active Comparator): Continuous positive airway pressure is a CPAP given at effective pressure to decrease the work of breathing in COPD patients
  Interventions: Device: continuous positive airway pressure

INTERVENTIONS:
Device: continuous positive airway pressure — positive airway pressure given by a medical device through a nasal mask

SUMMARY:
Static hyperinflation is frequent in Chronic obstructive pulmonary disease (COPD) , resulting in increased end expiratory lung volume and positive end expiratory pressure (PEEPi) at the end of a normal expiration.

Static hyperinflation worsens the work of breathing is increases patient's dyspnea.

The application of a continuous positive airway pressure (CPAP) has been shown to improve static hyperinflation and to decrease the work of breathing.

Sleep is deteriorated in COPD patients, and causal factors includes static hyperinflation. The purpose of our study is to assess the effect of nocturnal CPAP on sleep quality and functional respiratory parameters.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is characterized by an airflow obstruction, inducing a flow limitation. As a consequence, we observe in these patients an increased end expiratory lung volume and a positive end expiratory pressure (PEEPi) at the end of a normal expiration.

Patients are breathing at higher pulmonary volumes: this is the concept of static hyperinflation.

This worsens the breathing pattern because in this situation, the work of breathing is increased such that dyspnea increases.

The application of a continuous positive airway pressure (CPAP) has been shown to improve static hyperinflation and to decrease the work of breathing.

Sleep is deteriorated in COPD patients, and causal factors includes static hyperinflation, cough, depression. Moreover, normal physiological changes occuring during sleep in COPD patients are leading to deterioration of gaseous exchanges. The purpose of our study is to assess the effect of nocturnal CPAP on sleep quality and functional respiratory parameters.

ELIGIBILITY:
Inclusion Criteria:

* stable chronic obstructive pulmonary disease patients exhibiting a FEV1<80 %,

Exclusion Criteria:

* Known sleep apnea syndrome or other sleep disease interfering with sleep quality
* Body mass index > 30 kg/m2
* heart failure
* hypnotics intake

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
sleep quality | day 1
  sleep efficiency, total sleep time, sleep architecture measured by polysomnography

SECONDARY OUTCOMES:
static hyperinflation | day 1
  measure of static hyperinflation by lung function test after the night spent with CPAP

IPD SHARING:
Plan to Share IPD: No